CLINICAL TRIAL: NCT02014571
Title: A Randomized, Single Blind, Dose Escalation, Placebo-Controlled Study to Assess the Safety, Pharmacokinetics, and Antiviral Activity of Repeat Doses of GSK2878175 in Subjects With Chronic Hepatitis C.
Brief Title: Study to Assess the Safety, Pharmacokinetics, and Antiviral Activity of Repeat Doses of GSK2878175 in Subjects With Chronic Hepatitis C.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 116976
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis C, Chronic
Keywords: NS5B; chronic hepatitis C (CHC); antiviral activity; pharmacokinetics (PK); Safety; hepatitis C virus (HCV); GSK2878175
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — GSK2878175

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort A (Experimental): Eight subjects will be randomized to receive either 10 mg of GSK2878175 active treatment (4 HCV genotype 1a [GT1a] and 2 HCV genotype 1b [GT1b]) or matching placebo (1 GT1a and 1 GT1b) daily for 2 days fasted.
  Interventions: Drug: GSK2878175; Drug: Placebo
- Cohort B (Experimental): Eight subjects will be randomized to receive either 30 mg of GSK2878175 active treatment (4 GT1a and 2 GT1b) or matching placebo (1 GT1a and 1 GT1b) daily for 2 days fasted.
  Interventions: Drug: GSK2878175; Drug: Placebo
- Cohort C (Experimental): Eight subjects will be randomized to receive either GSK2878175 active treatment (4 GT1a and 2 GT1b) or matching placebo (1 GT1a and 1 GT1b) daily for 2 days fasted.
  Interventions: Drug: GSK2878175; Drug: Placebo
- Cohort D (Experimental): Twenty subjects will be randomized to receive either 60 mg of GSK2878175 active treatment (6 GT2, 6 GT3, 3 GT4) or matching placebo (2 GT2, 2 GT3, 1 GT4).
  Interventions: Drug: GSK2878175; Drug: Placebo

INTERVENTIONS:
Drug: GSK2878175 — Round tablets (5.0mg) given once daily repeated (to 2 days), oral dose.
Drug: Placebo — Round tablets (5.0mg) given once daily repeated (to 2 days), oral dose visually matching GSK2878175.

SUMMARY:
GSK2878175 is a site IV NS5B non-nucleoside inhibitor (NNI) being developed for the treatment of chronic hepatitis C virus (HCV) infection. The purpose of this study is to investigate the effects of GSK2878175, at different doses in men and women infected with chronic hepatitis C virus. The study will investigate how much of the drug gets into the blood stream and how long the body takes to get rid of it. The study will also investigate if GSK2878175 has any important side effects. The study will also measure what effect GSK2878175 has on the hepatitis C virus infection after taking the study medication for 2 days. Approximately 44 people will take part in this study. Depending on the type of chronic hepatitis C infection a subject will be enrolled into 1 of 4 groups randomly. Each group will participate in one dosing session. One dosing session consists of GSK2878175 or a placebo (sugar pill) given once per day for 2 days.

Group A, B, and C is made up of 8 participants per group. In each of these groups 6 participants will receive GSK2878175 and 2 participants will receive placebo. Group D is made up of 20 participants. 15 participants will receive GSK2878175 and 5 participants will receive placebo. The treatment groups will be dosed in sequence. Group A will be the first to take the study medication, then Group B, and so on. The plan is to dose subjects in Group A with 10 mg, Group B with 30 mg, Group C with 60 mg, and Group D with 60 mg of GSK2878175 or placebo. The next treatment group's actual dose will be decided after looking at the results from the previous group. The doses may therefore be higher or lower than planned depending on the previous group's results. The number of participants enrolled in the next group may also change depending on the results from the previous group.

ELIGIBILITY:
Inclusion Criteria:

* Has chronic genotype 1 (subtypes 1a or 1b) or genotype 2 or genotype 3 or genotype 4 (as assessed by VERSANT® HCV Genotype assay 2.0 (LiPA); VERSANT is a registered trademark of the Siemens Healthcare company.) HCV infection documented by at least 1 measurement of serum HCV RNA >=100,000 IU/mL measured during Screening by the COBAS® High Pure/COBAS TaqMan® HCV Test v2.0 (COBAS and TaqMan are registered trademarks of the Roche Molecular Diagnostics company.) and at least one of the following:

Documented HCV serology demonstrating the presence of anti-HCV antibodies at least 6 months before screening; or Documented presence of HCV RNA at least 6 months before screening; or Documented evidence of fibrosis on liver biopsy obtained within 3 years (<36 calendar months) prior to the Day 1visit; or FibroSure/FibroTest >0.28 and <=0.58 at screening (Note: subjects with a FibroTest score <=0.28 may be included as long as they meet any 1 of the other CHC criteria above).

Note: Cohorts are genotype specific.

* Agrees to IL28B genotyping.
* The subject is able to understand and is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form and is likely to complete the study as planned.
* Subjects must be treatment-naïve and have not received prior treatment with any interferon, immunomodulatory agent, or DAA for HCV.
* Male or female aged between 18 and 60 years of age, inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MIU/ml and estradiol <40 pg/ml (<147 pmol/L) is confirmatory].

Child-bearing potential with negative pregnancy test as determined by serum hCG test (at Screening and Day -1) and urine hCG test on Day 1 and:

Agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 28 days post last dose.

OR has only same-sex partners, when this is her preferred and usual lifestyle.

* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until the follow up visit (14 days post last dose).
* Body weight >50kg (110 lb) for men and >45kg (99 lb) women and a body mass index (BMI) between 18.5-35 kg/m^2 inclusive will be allowed.
* The subject's systolic blood pressure is inside the range of 90-140 mmHg, and diastolic blood pressure is inside the range of 45-90 mmHg. Heart rate is inside the range of 50-100 bpm for female subjects or 45-100 bpm for male subjects.
* Is otherwise healthy as determined by the medical history, physical examination, ECG findings, and clinical laboratory measurements performed at Screening.
* Aspartate transaminase (AST), Alanine transaminase (ALT), and Alkaline Phosphatase (ALP) <2X Upper Limit of Normal (ULN).
* Total bilirubin <2X ULN (except in subjects with Gilbert's syndrome).
* Absolute neutrophils count >=1000/mm^3.
* Albumin >=3.5 g/dL.
* Platelet count >=140000/mm^3.
* Hemoglobin:

>=11 g/dL for female subjects >=12 g/dL for male subjects Note: for subjects who have baseline hemoglobin below the lower limit of normal, attention should be paid to correctable causes of anemia such as iron, folate, or B12 deficiency.

* All other hematology and clinical chemistry; no clinically significant abnormalities or laboratory values that preclude treatment.
* Based on single or averaged QTc values of triplicate ECGs obtained over a brief recording period:

QTcF <450 msec; or QTcF <480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* History of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject.
* Family history of prolonged QT syndrome (Torsade de Pointes) or sudden cardiac death; first-degree relative with myocardial infarction at premature age (<=45 years for male relative; <=55 years for female relative).
* History or other clinical evidence of hypertension, significant or unstable cardiac disease (e.g., prolonged QT syndrome [torsade de pointes], angina, congestive heart failure, myocardial infarction, diastolic dysfunction, significant arrhythmia, coronary heart disease, and/or clinically significant ECG abnormalities).
* Evidence of cirrhosis, as determined by any 1 of the following:

FibroSure/FibroTest score >0.58; or Liver biopsy with a fibrosis stage indicative of cirrhosis as classified by a local pathologist (defined as Knodell >3, Metavir >2, Ishak >4, or Batts and Ludwig >2). Both incomplete and transition to cirrhosis (e.g., Metavir score 3) are considered as cirrhosis; or History of ascites, hepatic encephalopathy, or esophagogastric varices.

* Active malignant disease or history of malignant disease within 5 years before screening, with the exception of successfully treated basal cell carcinoma, squamous cell cancer of the skin, and carcinoma of the cervix in situ.
* Any other cause of significant liver disease in addition to hepatitis C, which may include but is not limited to malignancy with hepatic involvement, hepatitis B, druginduced or alcohol-related liver disease, autoimmune hepatitis, hemochromatosis, Wilson's disease, nonalcoholic steatohepatitis, or primary biliary cirrhosis.
* Estimated creatinine clearance ≤50 mL/min using the Cockcroft-Gault equation at screening.
* A medical condition that requires frequent or prolonged use of systemic corticosteroids or immunosuppressive drugs (e.g., severe asthma; severe arthritis or autoimmune conditions; organ transplantation; or acute adrenal insufficiency).
* History of regular alcohol consumption within 1 month of the study defined as:

an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.

* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice, pummelos, satsuma, ugli, tangerine, and tangelo, exotic citrus fruits, grapefruit hybrids or fruit juices from 5 days prior to the first dose of study medication.
* A positive pre-study Hepatitis B surface antigen result within 3 months of screening.
* A positive test for HIV antibody.
* A positive pre-study drug/alcohol screen. Unwilling to refrain from use of the illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* Holter monitoring shows one or more of the following:

Any symptomatic arrhythmia (except isolated extra systoles). Sustained cardiac arrhythmias (such as atrial fibrillation or flutter, SVT (>10 consecutive beats).

Sinus tachycardia (or supraventricular tachycardia) greater than 150 bpm. Non-sustained or sustained ventricular tachycardia (defined as >3 consecutive ventricular ectopic beats).

Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher in an awake subject], WPW syndrome, other pre-excitation syndromes).

Symptomatic sinus pause or sinus pause >3 seconds - unless subject is straining, vomiting, or having some other type of hypervagal response.

300 or more supraventricular ectopic beats in 24 hours. 250 or more ventricular ectopic beats in 24 hours. Ischemia, diagnosed by a sequence of ECG changes that include flat or down sloping ST-segment depression >0.1 mV, with a gradual onset and offset that lasts for a minimum period of 1 minute. Each episode of ischemia must be separated by a minimum duration of at least 1 minute, during which the ST segment returns back to baseline (1x1x1 rule).

* Unable to use spirometry equipment correctly.
* Abnormal spirometry results:

FEV1 less than 80% of predicted value FEV1/FVC less than 70%

* History of or active diagnosis of pulmonary disease such as asthma, emphysema, chronic obstructive pulmonary disease (COPD) or interstitial lung disease.
* History of or active diagnosis of thyroid disease.
* Any condition possibly affecting drug absorption (e.g., gastrectomy or other significant gastrointestinal tract surgery, such as gastroenterostomy, small bowel resection, or active enterostomy).
* Lactating females.
* Where participation in the study would result in donation of blood or blood products in excess of 550 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2013-12-26 (Actual); Primary Completion 2014-07-03 (Actual); Study Completion 2015-01-15 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by the collection of adverse events (AEs). | Screening to 14 days post last-dose
  AEs will be collected from the start of Study Treatment and until 14 days post last-dose (at follow up).
Safety as assessed by hematology, clinical chemistry, urinalysis, vital signs, electrocardiogram (ECG) intervals, ECG rhythm telemetry, pulmonary function tests, respiratory rate and lung auscultation. | Pre-dose to 14 days post last-dose
  Absolute values and changes over time of hematology, clinical chemistry, urinalysis, vital signs (blood pressure [BP], FSH/Estradiol (Women), Urine β-hCG (Women) temperature, and heart rate), 12 LED ECG, and Holter monitoring, ECG intervals, ECG rhythm, and telemetry will be measured. Telemetry is the continuous monitoring of a subject's heart rate and rhythm from a remote location. Pulmonary function testing includes a group of tests that measure how well the lung is functioning.
Composite of PK parameters (Day 1) following repeat dose administration of GSK2878175. | Pre Dose, 0.5hr, 1.5hr, 4hr, 6hr, 12hr
  PK parameters include: AUC (0-24), Tmax, Cmax,C24, t1/2, tlag, CL/F for Day 1
Composite of PK parameters (Day 2) following repeat dose administration of GSK2878175. | Day 2 Pre Doseand Post Day 1 Dose at 24hr, 24.5hr, 25.5hr, 28hr, 30hr, 33hr, 36hr, 48hr, 72hr, 96hr, 144hr, 192hr, 240hr and 360hr
  PK parameters include: AUC (0-t), Ct, Cmax, tmax, t1/2, CL/F for Day 2.
Antiviral activity as assessed by HCV RNA viral load. | Baseline, 24 hr, 48 hr, and 72 hr
  HCV RNA viral load reduction from baseline at the 24 hr, 48 hr, and 72 hr timepoints during dosing of GSK2878175 in HCV subjects
Antiviral activity as assessed by HCV RNA maximum change. | Pre-dose to 14 days post last-dose.
  HCV RNA change from baseline to nadir (maximum change) in CHC subjects.
Antiviral activity as assessed by Time course of HCV viral load. | Baseline, Day1, Day 2, Day 3, Day 4, Day 5, Day 7, Day 9, Day 11, and Day 16 (Follow Up Visit)
  Time course of HCV viral load at baseline, during, and after dosing with GSK2878175.

SECONDARY OUTCOMES:
Viral quasi-species population. | Pre Dose and 12hr on Day 1 and at 24hr, 30hr, 36hr, 48hr, 72hr, 96hr, 144hr, 192hr, 240hr and 360hr Post 1st Dose
  Sequence analysis of the viral quasispecies population as appropriate before and after a repeat dose.
IL28B rs12979860 status on GSK2878175 pharmacokinetics. | Day 1 Pre Dose.
  Determination of IL28B status (C/C versus carriage of the T allele) status on GSK2878175 pharmacokinetics or exposure-response relationship.
Exposure-response relationships for various safety parameters, if appropriate. | Pre-dose to 14 days post last-dose
  Correlation between PK parameters and various safety parameters, if appropriate.
Exposure-response relationship for antiviral effect. | 24, 48 and 72 hours after the first dose.
  Correlation between PK parameters and changes in HCV RNA viral load at 24, 48 and 72 hours after the first dose.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: Results for study 116976 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116976?search=study&study_ids=116976#rs